CLINICAL TRIAL: NCT00666796
Title: A Randomized, Double-Blind, 4-way Crossover, Placebo-Controlled, Single Center Trial to Evaluate the Potential Pharmacodynamic Interaction Between Gabapentin 500 mg and Ethanol in Healthy Volunteers
Brief Title: A Study to Assess the Pharmacodynamic Interaction Between Gabapentin and Ethanol in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: A9451149
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2008-04

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Ethanol; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Placebo Comparator)
  Interventions: Drug: Placebo ethanol; Drug: Placebo
- B (Experimental)
  Interventions: Drug: Ethanol; Drug: Gabapentin
- C (Experimental)
  Interventions: Drug: Ethanol; Drug: Placebo
- D (Experimental)
  Interventions: Drug: Gabapentin; Drug: Placebo ethanol

INTERVENTIONS:
Drug: Placebo ethanol — Matched placebo ethanol 0.4% in a total volume of 300 mL as an orange juice cocktail (consumed within 15 minutes) at 1 hour prior to assessment timepoint
  Arms: A
Drug: Ethanol — Ethanol 0.7 g/kg in a total volume of 300 mL as an orange juice cocktail (consumed within 15 minutes) at 1 hour prior to assessment timepoint
  Arms: B
Drug: Placebo — Matched placebo oral capsule with 8 oz of water 2 hours prior to assessment timepoint
  Arms: A
Drug: Gabapentin — Gabapentin 500 mg oral capsule with 8 oz of water 2 hours prior to assessment timepoint
  Arms: B
Drug: Ethanol — Ethanol 0.7 g/kg in a total volume of 300 mL as an orange juice cocktail (consumed within 15 minutes) at 1 hour prior to assessment timepoint
  Arms: C
Drug: Placebo — Matched placebo oral capsule with 8 oz of water 2 hours prior to assessment timepoint
  Arms: C
Drug: Gabapentin — Gabapentin 500 mg oral capsule with 8 oz of water 2 hours prior to assessment timepoint
  Arms: D
Drug: Placebo ethanol — Matched placebo ethanol 0.4% in a total volume of 300 mL as an orange juice cocktail (consumed within 15 minutes) at 1 hour prior to assessment timepoint
  Arms: D

SUMMARY:
The purpose of this study is to assess the pharmacodynamic interaction between gabapentin and ethanol

ELIGIBILITY:
Inclusion Criteria:

* Volunteers in good health aged 21 to 50 (inclusive) years who weigh 50 to 100 kg (110-220 lbs.)
* Experience with alcohol, defined as mild to moderate use of alcohol, ie, maximum of 14 alcoholic drinks per week

Exclusion Criteria:

* Recent history (within 2 years) of, or current treatment for, a sleeping disorder including excessive snoring, obstructive sleep apnea or a chronic painful condition
* Recent history (within 2 years) of, or clinical evidence of significant unstable or uncontrolled respiratory (including asthma and congestive obstructive pulmonary disease), cardiovascular, gastrointestinal, hepatic, renal, endocrine, neurologic (including seizures), psychiatric or other chronic disease
* History of alcoholism or drug abuse; recreational drug use within the past 30 days; use of benzodiazepines, Ambien®, Sonata®, antidepressants or psychoactive medication within 30 days prior to screening; use of any other sedative, hypnotic, antihistamine, anticholinergic, melatonin, DHEA or herbal sleep/relaxation remedy within 7 days prior to screening

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-04; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Change from pre-dose in the Psychomotor Vigilance Task (PVT) for completed subjects | 2 hours post-dose

SECONDARY OUTCOMES:
Change from pre-dose in DSST for Intent-to-Treat (ITTI subjects | 2 and 6 hours post-dose
Change from pre-dose in PVT for ITT subjects | 2 and 6 hours post-dose
Change from pre-dose in Buschke Selective Reminding Test (BSRT) for completed subjects | 2 and 6 hours post-dose
Change from pre-dose in BSRT for ITT subjects | 2 and 6 hours post-dose
Change from pre-dose in Stanford Sleepiness Scale (SSS) for completed subjects | 2, 6, and 7.5 hours post-dose
Change from pre-dose in SSS for ITT subjects | 2, 6, and 7.5 hours post-dose
Adverse events | Throughout study duration
Vital signs | Throughout study duration
Change from pre-dose in PVT for completed subjects | 6 hours post-dose
Change from pre-dose in Digit Symbol Substitution Test (DSST) for completed subjects | 2 and 6 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Miami, Florida, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9451149&StudyName=A%20Study%20to%20Assess%20the%20Pharmacodynamic%20Interaction%20between%20Gabapentin%20and%20Ethanol%20in%20Healthy%20Subjects